CLINICAL TRIAL: NCT06591221
Title: Evaluation of the Effectiveness of Manual Maintenance Therapy (Chuna Maintenance Therapy) for Chronic Bothersome Neck Pain : a Multi-centered, Pragmatic Randomized Controlled Study
Brief Title: The Effectiveness of Chuna Maintenance Therapy for Chronic Bothersome Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2024-02
Record Dates: First submitted 2024-08-31; First posted 2024-09-19 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Chronic Pain
Keywords: Chuna therapy; Manual therapy; Chronic neck pain
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chuna maintenance therapy group (Experimental): This group will receive chuna therapy determined by the clinician based on the subject's symptoms, degree of improvement, etc. (1 time/2 weeks, total 20 weeks)
  Interventions: Procedure: Chuna Maintenance Therapy
- Lifestyle management & self-exercise group (Other): This group will perform lifestyle management and daily self-exercise. The exercise education will be performed per 4 weeks for total 20 weeks.
  Interventions: Procedure: Chuna Maintenance Therapy

INTERVENTIONS:
Procedure: Chuna Maintenance Therapy — it is conducted every two weeks for a total of 20 weeks for individuals. The technique follows the guidelines of the Society of Chuna Manual Medicine and is based on Chuna Medicine (2.5th edition), which is utilized as a textbook in Korean Medicine colleges.
  The treatment is selectively administered based on the clinical judgment of the practitioner.

SUMMARY:
This study is a pragmatic randomized controlled study that assessed 250 subjects complaining of chronic bothersome neck pain with mild discomfort in a 1:1 ratio: chuna maintenance therapy group (125 subjects, 1 time/2 weeks, total 20 weeks) and lifestyle management & self-exercise group (125 subjects, exercise method education 1 time/4 weeks, total 20 weeks).

ELIGIBILITY:
* Inclusion Criteria:

  1. Aged 19 or older but under 70.
  2. Neck pain with pain duration of 12 months or longer
  3. NRS of neck pain over the past month is 2 or more but less than 4
  4. Patients who have agreed to trial participation and provided written informed consent
* Exclusion Criteria:

  1. Patients diagnosed with serious pathology(s) which may cause neck pain (e.g. spinal metastasis of tumor(s), acute fracture, spinal dislocation)
  2. Patients with progressive neurologic deficit or severe neurologic symptoms such as spinal cord injury
  3. Patients whose pain is due to soft tissue disease not the spine (e.g. tumors, fibromyalgia, rheumatoid arthritis, gout)
  4. Patients with other chronic disease(s) which may interfere with treatment effect, safety, or interpretation of outcome (e.g. stroke and myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy)
  5. Patients currently taking steroids, immunosuppressants, medicine for mental illness or other medication(s) that may interfere with study results
  6. Pregnant patients or patients with plans of pregnancy or lactating patients
  7. Patients within 3 months after cervical surgery
  8. Patients with experience of participating in another clinical study within 1 month or plan to participate in another clinical study during the study participation and follow-up period within 6 months from the participation date
  9. Patients having difficult to completing the written informed consent
  10. Patients who are deemed unsuitable by the researchers

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NRS (Numeric rating scale) | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
  Ranging 0-10 likert scale (higher=worse)
NDI (Neck disability index) | Wk 1, 5, 9, 13, 17, 21, 25
  Each of the 10 items scores from 0 to 5, The maximum score is 50 (higher=worse)

SECONDARY OUTCOMES:
VAS(Visual analogue scale) for pain | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
  Ranging 0-10cm scale (higher=worse)
Number of days with bothersome neck pain | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
Recurrence | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
PGIC (Patient Global Impression of Change) | Wk 21, 25
  PGIC is a 7 point scale depicting a patient's rating of overall improvement (higher=worse)
EQ-5D-5L( The 5-level EuroQol-5) | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
  5 items for self-rating of overall health (lower=worse)
HINT-8 (health-related quality of life instrument-8) | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
  8 items for self-rating of overall health (lower=worse)
Rating for Credibility and Expectancy of the treatment | Once at screening procedure
  Ranging 1-9 likert scale (higher=more credible, positive results are expected)
Drug consumption history | Wk 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 25
  Whether medication was used (Y/N)

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon
  - Haeundae Jaseng Hospital of Korean Medicine, Haeundae
  - College of Korean Medicine, Kyung Hee University, Seoul
  - Department of Acupuncture & Moxibustion Medicine, College of Korean Medicine, Kyung Hee University, Seoul
  - Jaseng Hospital of Korean Medicine, Seoul
  - School of Korean Medicine, Pusan National University, Yangsan

IPD SHARING:
Plan to Share IPD: No